CLINICAL TRIAL: NCT00140621
Title: A Multicenter Open-label Study of the Safety and Efficacy of α-galactosidase A (R-h α-GAL) Replacement Therapy in Patients With Cardiac Fabry Disease
Brief Title: A Safety and Efficacy Study of Fabrazyme® Replacement Therapy in Patients With Cardiac Fabry Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGAL03204
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Results first posted 2015-04-15 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-04

CONDITIONS: Fabry Disease
Keywords: cardiac fabry disease
MeSH Terms: conditions — Fabry Disease | interventions — agalsidase beta

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Agalsidase Beta (Experimental): Agalsidase beta 1 milligram per kilogram (mg/kg) intravenously once every 2 weeks up to 156 weeks.
  Interventions: Drug: Agalsidase beta

INTERVENTIONS:
Drug: Agalsidase beta
  Other Names: Fabrazyme®

SUMMARY:
This is a multi-center, open label, phase IV study conducted to evaluate the efficacy and safety of agalsidase beta (Fabrazyme [recombinant form]) administered by intravenous drip infusion in participants with cardiac Fabry disease.

Participants participated for 4 weeks or less in the baseline period and 156 weeks for the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Participants definitively diagnosed with cardiac Fabry disease (who fulfill all of the following criteria)

  * In the case of male participants, documented plasma or leukocyte alpha-galactosidase A (α-GAL) activity was no more than 20 percent (%) of normal value (except for heterozygous female participants)
  * Left ventricular hypertrophy was noted.
  * Accumulation of globotriaosylceramide (GL-3) in the myocardium or a genetic deficiency associated with α-GAL was confirmed
  * Or in the case of heterozygous female participants, when the family (father or son) was diagnosed with Fabry disease. (Father or son was related by birth.)
  * Without symptoms or signs of Fabry, such as acroparesthesia, angiokeratomas, abnormal sweating, pain of distal extremities, chronic abdominal pain/diarrhea and corneal opacities were observed, except for proteinuria sign.
* Participants with interventricular and posterior wall thickness of at least 13 millimeter (mm) on echocardiography within 3 months before signed date to informed consent
* Participants in whom cardiac function was rated as Class I or II according to the New York Heart Association (NYHA) classification when giving informed consent.
* Participants classification: inpatients and outpatients
* Participants who had given written informed consent before the study-related baseline tests.

Exclusion Criteria:

* Participants with severe hypertension (for example, blood pressure more than or equal to 180 millimeter of mercury [mmHg] and/or blood pressure more than or equal to 110 mmHg in spite of adequate medication)
* Participants whose serum creatinine level was higher than the upper normal limit within 3 months (12 weeks) prior to giving informed consent.
* Participants who had undergone kidney transplantation or were currently on dialysis.
* Participants with any serious hepatic disorder. Participants who had abnormal hepatic function test values within 3 months (12 weeks) prior to giving informed consent (when either alanine aminotransferase [ALT] or aspartate aminotransferase [AST] level exceeded the value five times as high as the upper normal limit).
* Permanent pacemaker or defibrillator implanted participants
* Pregnant or lactating women
* Participants who had taken this drug for 6 months (26 weeks) or more before giving informed consent.
* Participants who had participated in a clinical study employing any other investigational product within 3 months prior to giving informed consent.
* Enzyme replacement therapy history, except for agalsidase beta
* Participants who were unwilling to comply with the requirements of the protocol.
* Others judged by the investigator or sub-investigator to be ineligible for the study

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2005-07; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (7):
- Japan (7):
  - Fujita Health University Hospital, Aichi
  - Sapporo Medical University Hospital, Hokkaido
  - Akune Citizen Hospital, Kagoshima
  - Tohoku University Hospital, Miyagi
  - Nihon University Itabashi Hospital, Tokyo
  - Nihon University Nerima Hikarigaoka Hospital, Tokyo
  - Yamanashi Prefectural Central Hospital, Yamanashi

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 7 centers between July 06, 2005 and August 6, 2012. One participant was treated at 2 study sites because the participant had to be transferred to another site during the study.
Groups:
- Agalsidase Beta (Fabrazyme [Recombinant Form]): Agalsidase beta 1 milligram per kilogram (mg/kg) intravenously once every 2 weeks up to 156 weeks.
Period: Overall Study
Arm/Group | Agalsidase Beta (Fabrazyme [Recombinant Form])
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Efficacy evaluable population (EEP) included all registered participants except those who had serious deviations from protocol compliance requirements, did not receive study drug, had no data available at baseline or after study drug administration, and who were found to have no condition in cardiac Fabry disease.
Groups:
- Agalsidase Beta: Agalsidase beta 1 mg/kg intravenously once every 2 weeks up to 156 weeks.
Arm/Group | Agalsidase Beta
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 1
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 58.50 (9.24)
Height [Mean (Standard Deviation); unit: centimeters (cm)] | 156.63 (7.20)
Left Ventricular Hypertrophy [Number; unit: participants]
  No | 0
  Yes | 6
Globotriaosylceramide (GL-3) Accumulation in the Myocardium [Number; unit: participants]
  No | 0
  Yes | 1
  Not Measured | 5

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Interventricular Septum and Left Ventricular Posterior Wall Thickness at Week 156
Description: Interventricular septum and left ventricular posterior wall thickness was assessed by echocardiogram.
Time Frame: Baseline to Week 156
Population: EEP.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Groups:
- Agalsidase Beta: Agalsidase beta 1 mg/kg once every 2 weeks as an intravenous infusion up to 156 weeks.
Arm/Group | Agalsidase Beta
Number analyzed (Participants) | 6
percent change
  Interventricular septum wall thickness | -3.31 [-19.67 to 16.39]
  Left ventricular posterior wall thickness | -6.34 [-21.47 to 11.71]

2. Primary Outcome: Change From Baseline in Interventricular Septum and Left Ventricular Posterior Wall Thickness at Week 156
Description: Interventricular septum and left ventricular posterior wall thickness was assessed by echocardiogram.
Time Frame: Baseline to Week 156
Population: EEP.
Measure: Least Squares Mean (95% Confidence Interval); unit: mm
Arm/Group | Agalsidase Beta
Number analyzed (Participants) | 6
mm
  Interventricular septum wall thickness | 0.37 [-3.88 to 4.61]
  Left ventricular posterior wall thickness | -0.33 [-3.31 to 2.64]

3. Secondary Outcome: Number of Participants in Overall Cardiac Function Assessment and Clinical Symptoms at Week 156: Change From Baseline in Cardiac Function Test
Description: Overall cardiac function assessment was assessed by tests (echocardiogram,cardiac catheterization (optional),electrocardiogram,B-type natriuretic peptide [BNP]), clinical symptoms (subjective symptoms) and the New York Heart Association (NYHA) cardiac functional classification.Overall assessment of cardiac function was assessed based on the evaluation items including interventricular septum thickness, left ventricular posterior wall thickness, left ventricular mass, clinical function tests and clinical symptoms. A subject was considered to be Improved: if Improved in 2 items or more, Unchanged: Improved in one item and unchanged in 2 items or unchanged in all 3 items, Aggravated: Aggravated in one item or more.
Time Frame: Baseline to Week 156
Population: EEP.
Measure: Number; unit: participants
Arm/Group | Agalsidase Beta
Number analyzed (Participants) | 6
participants
  Improved | 5
  Unchanged | 0
  Aggravated | 1

4. Secondary Outcome: Percent Change From Baseline in GL-3 Plasma Levels at Week 156
Time Frame: Baseline to Week 156
Population: EEP.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Agalsidase Beta
Number analyzed (Participants) | 6
percent change | -18.91 [-42.35 to 14.07]

5. Secondary Outcome: Change From Baseline in Short Form (36) Health Survey (SF-36) Scores at Week 156
Description: The 36-Item Short-Form Health Survey (SF-36) is a standardized survey evaluating 8 aspects of functional health and well-being: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. These 8 aspects can also be summarized as physical component score (PCS) and mental component score (MCS). The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning).
Time Frame: Baseline to Week 156
Population: EEP.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Agalsidase Beta
Number analyzed (Participants) | 6
units on a scale
  Physical Health: PCS | 6.868 (15.238)
  Mental Health: MCS | 4.380 (7.425)

6. Primary Outcome: Percent Change From Baseline in Left Ventricular Mass (LVM) at Week 156
Description: Left ventricular mass was assessed by echocardiogram.
Time Frame: Baseline to Week 156
Population: EEP.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Agalsidase Beta
Number analyzed (Participants) | 6
percent change | -4.14 [-24.35 to 21.47]

7. Primary Outcome: Change From Baseline in LVM at Week 156
Description: Left ventricular mass was assessed by echocardiogram.
Time Frame: Baseline to Week 156
Population: EEP.
Measure: Least Squares Mean (95% Confidence Interval); unit: gm
Arm/Group | Agalsidase Beta
Number analyzed (Participants) | 6
gm | 22.70 [-106.57 to 151.97]

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from signature of the informed consent form up to the final visit (Week 156) regardless of seriousness or relationship to investigational product.
Description: Reported adverse events are treatment-emergent adverse events that is AEs that developed/worsened during the 'on treatment period' (from the first study infusion up to Week 156).
Arm/Group | Agalsidase Beta
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Agalsidase Beta (N=6)
Large intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Agalsidase Beta (N=6)
Nasopharyngitis (Infections and infestations) | 5
Chronic sinusitis (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Large intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1
Anxiety disorder (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 1
Middle insomnia (Psychiatric disorders) | 1
Headache (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 1
Intercostal neuralgia (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Palpitations (Cardiac disorders) | 4
Atrial fibrillation (Cardiac disorders) | 1
Atrioventricular block (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Bundle branch block right (Cardiac disorders) | 1
Left ventricular hypertrophy (Cardiac disorders) | 1
Supraventricular extrasystoles (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Ventricular hypertrophy (Cardiac disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Colonic polyp (Gastrointestinal disorders) | 1
Dental caries (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Gastritis erosive (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Oedema (General disorders) | 2
Chest discomfort (General disorders) | 1
Chest pain (General disorders) | 1
Chills (General disorders) | 1
Feeling hot (General disorders) | 1
Injection site inflammation (General disorders) | 1
Puncture site haemorrhage (General disorders) | 1
Tenderness (General disorders) | 1
Aspartate aminotransferase increased (Investigations) | 2
Alanine aminotransferase increased (Investigations) | 1
Blood pressure decreased (Investigations) | 1
Blood urea increased (Investigations) | 1
Body temperature decreased (Investigations) | 1
Heart rate increased (Investigations) | 1
Occult blood (Investigations) | 1
Protein urine present (Investigations) | 1
White blood cell count decreased (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to publishing results from this study in academic meetings, medical journals, etc., the investigator and subinvestigator of the post-manufacturing/marketing clinical study must obtain the approval from the sponsor of the post-manufacturing/marketing clinical study in writing.